CLINICAL TRIAL: NCT04055571
Title: Evaluation of Outcomes From Treatment of Benign or Malignant Pancreatic Diseases
Status: Recruiting | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 036.HPB.2018.R
Record Dates: First submitted 2019-03-22; First posted 2019-08-13 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Benign or Malignant Pancreatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will be a retrospective chart review of patients who have been diagnosed with the benign or malignant pancreatic disease under the practice of Dr. Rohan Jeyarajah, M.D., Dr. Houssam Osman M.D., and Dr. Edward Cho M.D., Sc.M. at Methodist Health System Hospital in Richardson, TX. The investigators plan to conduct an analysis of patients meeting the inclusion criteria from 2005 to present. Study will also be conducted by the PI, Sub-Is, surgery fellows, office staff and clinical research coordinator who are delegated to do by the PI. Data will be obtained by looking through either investigator's patients or through a national database. Data will be analyzed primarily by the study conductors.

DETAILED DESCRIPTION:
It is reported in the literature that the treatment of any pancreatic disease process, whether benign or malignant, continues to be a huge challenge. For example, patients with adenocarcinoma continue to be diagnosed at an advanced stage with medical and surgical options that are improving in terms of outcome measurements but with much more room for improvement. The investigator's goal is to continue to review our treatment outcomes to further improve overall survival, overall symptom control, mortality, and morbidity.

The main aim of this study is to evaluate and compare the outcomes from the investigator's decisions on multiple treatments of benign or malignant pancreatic diseases.There is a need to understand and improve the current diagnosis and treatment algorithm for pancreatic pathologies. Continued evaluation and study is imperative to ensure that national guidelines are improving to enhance patient cure and/or recovery.

All past patients who were treated for a particular benign or malignant pancreatic disease process under evaluation from 2005 to present will be included in this study.

ELIGIBILITY:
Inclusion Criteria:

* • All patients diagnosed and treated for pancreatic diseases, benign or malignant from 2005 to present

  * Age ≥18 years

Exclusion Criteria:

* • Patients that are not diagnosed with or treated for pancreatic diseases

  * Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All past patients who were treated for a particular benign or malignant pancreatic disease process under evaluation from 2005 to present will be included in this study.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-03-05 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2005 to 2019
  Number of patients who have been diagnosed with benign or malignant pancreatic disease

CONTACTS AND LOCATIONS:
Overall Officials: Dhiresh Jeyarajah, M.D., Principal Investigator — Methodist Richardson Medical Center
Locations (1):
- Trinity Surgical Consultants, Methodist Richardson Medical Center, Richardson, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Only de-identified PHI will be shared in relevant research mediums.